CLINICAL TRIAL: NCT04066673
Title: Intelligence Quotient Assessment in Children With Autistic Spectrum Disorders.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Mohammed Tawfeek, Resident of pediatric Department,, Assiut University
Other Study IDs: IQ in Autism
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stanford-Binet Intelligence Scale, 5th Edition — The SB5 is a descendent of the very first intelligence measure ever created. It tests general intellectual ability, and the Fifth Edition affords the ability to report Full Scale, Abbreviated, Nonverbal, and Verbal IQ scores

SUMMARY:
The aim of this study is to assess the cognitive strengths and weaknesses of children with autism and the possible effect of age and IQ on Stanford-Binet Intelligence Scale, 5th Edition. Such analysis will help us for prompt and early intervention.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASDs) are characterized by deficits in both social interaction and communication, as well as by restricted and repetitive patterns of behavior, and are a type of Pervasive Developmental Disorder (PDD). Intellectual disability (ID) is characterized by deficits in adaptive functioning, an intelligence quotient (IQ) that falls at least two standard deviations below average (i.e., below 70), and onset prior to adulthood (American Psychiatric Association, 2000).

Although ID is not a core symptom of ASD, there is an established relationship between the two constructs. Seventy percent of children with AD have a co-morbid diagnosis of ID (Bolte & Poustka, 2002; Fombonne, 2005). It has been suggested that many children who would have been diagnosed with ID in the past would today receive an ASD diagnosis, even with identical symptomatology (Lecavalier et al., in press).

The SB5 is a descendent of the very first intelligence measure ever created. It tests general intellectual ability, and the Fifth Edition affords the ability to report Full Scale, Abbreviated, Nonverbal, and Verbal IQ scores(Roid, 2003).. One of the updated features of the SB5 is the nonverbal component, in that close to half of the responses no longer require verbal answers (Coolican, Bryson & Zwaigenbaum, 2008).The Full Scale IQ is derived from the verbal and nonverbal scales, each with five subtests bearing the same names: Fluid Reasoning, Knowledge, Quantitative Reasoning, Visual Spatial Processing, and Working Memory.

ELIGIBILITY:
Inclusion Criteria:

* Age: from3 to18 years
* Gender: both sexes will be included in the study
* Clinical ASD diagnosis.
* Full Scale test results available for SB5.

Exclusion Criteria:

* 1- Age below 3years or above 18 years. 2- Mental Retardation due to other causes than autism. 3- Presence of other chronic illnesses affecting their quality of lives.

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Forty children will participate in the study, clinically diagnosed by CARS Scoring IQ will be assessed by Stanford-Binet Intelligence Scales, 5th Edition have autism .They will be recruited from children attending Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Intelligence Quotient assessment in autistic children by the Stanford-Binet Intelligence Scales, 5th Edition | Baseline
  assess the cognitive strengths and weaknesses of children with autism and the possible effect of age and IQ on Stanford-Binet Intelligence Scale, 5th Edition.

REFERENCES:
- [Background] Bolte S, Poustka F. The relation between general cognitive level and adaptive behavior domains in individuals with autism with and without co-morbid mental retardation. Child Psychiatry Hum Dev. 2002 Winter;33(2):165-72. doi: 10.1023/a:1020734325815. PMID 12462353
- [Background] Coolican J, Bryson SE, Zwaigenbaum L. Brief report: data on the Stanford-Binet Intelligence Scales (5th ed.) in children with autism spectrum disorder. J Autism Dev Disord. 2008 Jan;38(1):190-7. doi: 10.1007/s10803-007-0368-2. Epub 2007 Apr 5. PMID 17410416